CLINICAL TRIAL: NCT06831838
Title: A Randomized Controlled Trial (RCT) to Determine the Efficacy of a Multidisciplinary CBT Based Pain Management Program for the Treatment of Aromatase Inhibitor Associated Musculoskeletal Symptoms (AIMSS) in Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-011941; NCI-2025-01395 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-02-11; First posted 2025-02-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Subjects randomized to the treatment group will participate in a multicomponent pain treatment program in addition to standard of care treatment.
  Interventions: Behavioral: Cognitive Behavioral Therapy based Pain Management Program
- Control Group (No Intervention): Subjects randomized to the control group will continue to receive standard of care treatment. At the end of the study, the control group participants will be offered the multicomponent pain treatment program.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy based Pain Management Program — Subjects will participate in a two-day structured class that will focus on Cognitive-Behavioral skills and strategies to improve pain control, fatigue, sleep disturbance, cognitive symptoms, and stress while educating patients on the efficacy of Aromatase Inhibitors in prolonging cancer-free survival with the goal of eliminating non-adherence.
  Arms: Treatment Group

SUMMARY:
The purpose of this research is to evaluate the effectiveness of a multidisciplinary pain management program for AIMSS in reducing pain, subjective cognitive complaints, psychological distress, and impaired functional status resulting in improved adherence to Aromatase Inhibitor medications compared to usual care. We want to identify predictors of improvement in pain, functional status, subjective cognition and mood following participation in the program.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* ECOG ≤ 2
* Stage 0-III HR+ breast cancer in need of strategies to reduce symptoms and improve quality of life

Exclusion Criteria:

• Less than 18 years of age.

- Stage 4 HR+ breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to Aromatase Inhibitors (AIs) | Baseline, 3 months, 6 months
  Adherence to Aromatase Inhibitors (AIs) medications will be collected as a self-reported question asking the patients if they have taken their medications as prescribed during the past month (yes vs. no).
AIMSS Follow-up Questionnaire | Baseline, 3 months, 6 months
  Subjects will complete the study follow-up questionnaire with study staff to indicate whether they are adhering to medications and to report symptoms.

SECONDARY OUTCOMES:
Brief Pain Inventory | Baseline, 3 months, 6 months
  The Brief Pain Inventory (BPI) allows participants to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. Possible scores range from 0 to 10 with higher scores indicating a worse outcome/more severe pain and interference.
Center for Epidemiologic Studies of Depression - Revised Questionnaire | Baseline, 3 months, 6 months
  The Center for Epidemiologic Studies Depression Scale-Revised (CESD-R) is a 20-item, self-reported questionnaire, that measures symptoms of depression. Each item is rated on a Likert scale, with 0 = 'Not at all or less than one day", and 3 = "Nearly every day for 2 weeks". Scores range from 0-60, with a score of 16 or higher indicating a risk of clinical depression.
Pain Catastrophizing Scale | Baseline, 3 months, 6 months
  he Pain Catastrophizing Scale (PCS) is a 13-item self-report measure designed to assess catastrophic thinking related to pain. Items are rated on 5-point Likert scale, with 0 = "Not at all" and 4 = "All the time" Higher score indicates higher level of catastrophizing.
Brief Resilience Scale | Baseline, 3 months, 6 months
  The Brief Resilience Scale is a 6 item, self-reported questionnaire, measuring how well a person recovers from stress. Each item is rated on a Likert scale, with 1 = "Strongly Disagree" and 5 = "Strongly Agree". The Brief Resilience Scale is scored by adding the value of all responses and dividing by 6. Higher scores indicate higher resilience to stress.
Social Support Survey | Baseline, 3 months, 6 months
  The Social Support Survey is a 4 item, self-reported questionnaire, assessing the availability of support. Items are rated on a 4 point Likert scale, with 0 = "None of the time" and 4 = "All of the time". Higher scores indicate a greater level of support.
World Health Organization (WHO) Disability Assessment Schedule | Baseline, 3 months, 6 months
  The WHO Disability Assessment Schedule is a 36-item, self-reported questionnaire, assessing health and disability. The questionnaire cover 6 domains: cognition, mobility, self-care, getting along, life activities, and participation. Each item is rated on a 5 point Likert scale, with 0 = "None" and 4 = "Extreme or Cannot do". Higher scores indicate greater disability.
State-Trait Inventory | Baseline, 3 months, 6 months
  The State-Trait Inventory is a self-reported questionnaire, used to assess anxiety. Participants respond to 40 questions about how they are currently feeling on a scale of 1 "Not at all" to 4 "Very much so". Total possible scores range from 40 to 160. Higher scores indicate higher anxiety (a worse outcome) and lower scores indicate less anxiety (a better outcome).
Cognitive Functioning Index (CFI) | Baseline, 3 months, 6 months
  The Cognitive Function Index (CFI) is a 14-item, self-reported questionnaire, used to assess cognitive status. Total scores range from 0-29, with higher scores indicating an increased perception about cognitive difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bruce, Ph.D., LP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials